CLINICAL TRIAL: NCT03116711
Title: Effects of Diet Type Selection Based on Response to a Carbohydrate Intolerance Questionnaire and Genetic Screening on Success to a Weight Loss and Exercise Program
Brief Title: Effects of Diet Selection Based on Genetic Screening on Success to a Weight Loss Program
Acronym: Curves3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Curves International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB2013-0737F
Record Dates: First submitted 2017-03-29; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Diet Modification
MeSH Terms: interventions — Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Positive CIQ plus High Carbohydrate Diet (Active Comparator): Positive Carbohydrate Intolerance Questionnaire (CIQ) plus 30% carbohydrate, 45% protein, 25% fat diet
  Interventions: Other: Positive CIQ plus High Carbohydrate Diet
- Positive CIQ plus High Protein Diet (Active Comparator): Positive Carbohydrate Intolerance Questionnaire (CIQ) plus 20% carbohydrate, 45% protein, 35% fat diet
  Interventions: Other: Positive CIQ plus High Protein Diet
- Negative CIQ plus High Carbohydrate Diet (Active Comparator): Negative Carbohydrate Intolerance Questionnaire (CIQ) plus 30% carbohydrate, 45% protein, 25% fat diet
  Interventions: Other: Negative CIQ plus High Carbohydrate Diet
- Negative CIQ plus High Protein Diet (Active Comparator): Negative Carbohydrate Intolerance Questionnaire (CIQ) plus 20% carbohydrate, 45% protein, 35% fat diet
  Interventions: Other: Negative CIQ plus High Protein Diet

INTERVENTIONS:
Other: Positive CIQ plus High Carbohydrate Diet — Positive Carbohydrate Intolerance Questionnaire plus High Carbohydrate Diet
  Arms: Positive CIQ plus High Carbohydrate Diet
Other: Positive CIQ plus High Protein Diet — Positive Carbohydrate Intolerance Questionnaire plus High Protein Diet
  Arms: Positive CIQ plus High Protein Diet
Other: Negative CIQ plus High Carbohydrate Diet — Negative Carbohydrate Intolerance Questionnaire plus High Carbohydrate Diet
  Arms: Negative CIQ plus High Carbohydrate Diet
Other: Negative CIQ plus High Protein Diet — Negative Carbohydrate Intolerance Questionnaire plus High Protein Diet
  Arms: Negative CIQ plus High Protein Diet

SUMMARY:
The purpose of this study is to determine the effects of diet type selection based on response to a Carbohydrate Intolerance Questionnaire (CIQ) and genetic screening on success to a weight loss and exercise program.

DETAILED DESCRIPTION:
The purpose of this study is to determine if stratification of individuals based on responses to a Carbohydrate Intolerance Questionnaire (CIQ), genetic screening, and/or DNA methylation affects weight loss success and/or health outcomes of women following the Curves moderate carbohydrate, high protein, low fat diet (30% carbohydrate, 45% protein, 25% fat) or the Curves carbohydrate restricted, high protein, moderate fat diet (20% carbohydrate, 45% protein, 35% fat).

ELIGIBILITY:
Inclusion Criteria:

* The participant is an apparently healthy female
* The participant is between the ages of 18 and 60

Exclusion Criteria:

* The participant is pregnant or nursing, or plans to become pregnant during the next 12 months or has been pregnant in the past 12 months
* The participant has uncontrolled metabolic disorder including known electrolyte abnormalities; heart disease, arrhythmias, diabetes, thyroid disease, or hypogonadism; a history of hypertension, hepatorenal, musculoskeletal, autoimmune, or neurological disease
* The participant is currently taking thyroid, hyperlipidemic, hypoglycemic, anti-hypertensive, or androgenic medications
* The participant has taken ergogenic levels of nutritional supplements that may affect muscle mass (e.g., creatine, HMB), anabolic/catabolic hormone levels (androstenedione, DHEA, etc.) or weight loss (e.g., ephedra, thermogenics, etc.) within the past three months
* The participant is willing to take participate in a regular moderate exercise program

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The eligibility criteria were at the request of the study sponsor.
Enrollment: 51 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Effects of diet selection on physical activity patterns changes (steps per day) | 24 weeks
Effects of diet selection on body weight changes (pounds) | 24 weeks
Effects of diet selection on hip/waist ratio changes (inches) | 24 weeks
Effects of diet selection on Resting Energy Expenditure (REE) changes (calories per day) | 24 weeks
Effects of diet selection on Blood Pressure (BP) changes (mmHG) | 24 weeks
Effects of diet selection on Heart Rate (HR) changes (beats per minute) | 24 weeks
Effects of diet selection on body composition (DXA) changes (percent fat mass) | 24 weeks
Effects of diet selection on Bioelectrical Impedance Analysis (BIA) changes (flow impedance) | 24 weeks
Effects of diet selection on a chemistry-15 blood panel changes | 24 weeks
Effects of diet selection on a cell blood count (CBC) blood panel changes | 24 weeks
Effects of diet selection on lipid panel changes | 24 weeks

SECONDARY OUTCOMES:
Effects of diet selection on maximal cardiopulmonary capacity changes (ml/kg/min) | 24 weeks
Effects of diet selection on muscular strength through a 1 repetition maximum (1 RM) test | 24 weeks
Effects of diet selection on muscular endurance through a maximal repetition test | 24 weeks
Effects of diet selection on gene expression changes | 24 weeks
Effects of diet selection on DNA methylation changes | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University

IPD SHARING:
Plan to Share IPD: No